CLINICAL TRIAL: NCT05906056
Title: Program of Continuous Passive Motion Exercises Against Heterotopic Ossification
Brief Title: Continuous Passive Motion Versus Heterotopic Ossification
Acronym: CPMversusHO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Professor of Phyical and Rehabilitation Medicine, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CPMUIoannina
Record Dates: First submitted 2023-05-08; First posted 2023-06-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Traumatic Brain Injury; Spinal Cord Injuries; Stroke
Keywords: Ossification, Heterotopic; continuous passive motion (CPM); zoledronic acid; range of motion (ROM); PROPHYLAXIS
MeSH Terms: conditions — Brain Injuries, Traumatic; Spinal Cord Injuries; Stroke; Ossification, Heterotopic | interventions — Motion Therapy, Continuous Passive; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Outcomes Assessor
Masking Description: CT will not reveal the group of patient's origin to the reader
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous passive motion (CPM) (Experimental): 10 ICU patients receiving CPM at HO joints that continuously stretches slowly the joint passively at a constant velocity in a painless range and for a substantial amount of time until there is evidence both laboratory (bone alkaline phosphatase) and radiographically (CT), that osteogenesis has entered a quiescent state. Conventional PT will also be performed.
  Plus a single dose of zoledronic acid (Aclasta) once the diagnosis of HO is made.
  Interventions: Device: Continuous Passive Motion (CPM); Other: Conventional physiotherapy (PT); Drug: Zoledronic Acid Injection
- Physiotherapy (PT) (Active Comparator): 10 ICU patients receiving the conventional PT, plus a single dose of zoledronic acid (Aclasta) once the diagnosis of HO is made.
  Interventions: Other: Conventional physiotherapy (PT); Drug: Zoledronic Acid Injection

INTERVENTIONS:
Device: Continuous Passive Motion (CPM) — CPM uses machines to move a joint passively i.e. without the patient exerting any effort. A motorized device moves the joint repetitively to a set of degrees and movement speed, determined by the caregiver either a medical doctor (physiatrist or orthopedic surgeon) or a physiotherapist. Its action preserves the joint's range of motion (ROM)
  Arms: Continuous passive motion (CPM)
Other: Conventional physiotherapy (PT) — Daily passive range of motion exercises (ROM) performed by the physiotherapist of the intensive care unit (ICU)
Drug: Zoledronic Acid Injection — one dose of intravenous zoledronic acid will be administered

SUMMARY:
The investigators hypothesize that Heterotopic Ossification (HO) formation can be suppressed if the application of a Continuous Passive Motion (CPM) device can be performed for a substantial amount of time. The investigators will use the following study design: a pilot study with 10 ICU patients receiving CPM and 10 matched cases which will follow a conventional physiotherapy program at the time of the conduction of the study. The comparison between the treatment and referent groups of the outcomes will prove the prophylactic power of CPM against HO.

DETAILED DESCRIPTION:
The aim of this study is to formally evaluate whether the investigators can indeed prevent HO by the timely and painless use of CPM in neurogenic intensive care unit (ICU) patients with stabilized medical conditions, suffering from neurological insults either traumatic brain injury (TBI), stroke, or Spinal Cord Injury (SCI). The investigators hypothesize that HO formation can be suppressed if CPM can be performed for a substantial amount of time. The investigators will perform a pilot study with 10 ICU patients receiving CPM and 10 matched cases which will follow a conventional physiotherapy program at the time of the conduction of the study. The primary outcomes will be the CT appearance of HO in the hip or knee joint and the degree of ROM limitation in the given joint at baseline and at the end of the clinical trial. A secondary outcome that will be measured, will be the Glasgow Coma Scale (GCS) at the beginning and at the end of the CPM program. The comparison between the treatment and referent groups in terms of these outcomes will prove the prophylactic power of CPM against HO.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stabilized medical condition suffering from neurological insult either traumatic brain injury (TBI), stroke, or Spinal Cord Injury.
2. A negative triplex ultrasound in order to rule out deep venous thrombosis (DVT)
3. A positive three-phase bone scan with Tc99. (Will be obtained as soon as HO symptoms are onset.)
4. Patients with verified HO formation on the knee or hip joint will undergo a CT to show the extent of the lesion.

Exclusion Criteria:

1. Life-threatening conditions that render Continuous passive motion (CPM) application difficult.
2. HO detected in another location than the hip or knee joint.
3. Concomitantly presence of other fractures that will interfere with the bone alkaline phosphatase (AP) level.
4. Patients not reacting to painful stimuli

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
ROM lost during the trial | According to the literature it is estimated to last approx. 70 days
  The difference in ROM between the measurements at baseline and at the end of the The program will last until there is evidence by CT and laboratory measurements (bone Alkaline Phosphatase) that osteogenesis has entered a quiescent state. prophylactic program
HO appearance on CT | According to the literature it is estimated to last approx. 70 days
  Based on Brooker HO classification method (between I and IV with IV being bridging bone and joint ankylosis), the difference in CT appearance at baseline and at the end of the program will serve as a descriptive tool. Until there is evidence by CT and laboratory measurements (bone Alkaline Phosphatase) that osteogenesis has entered a quiescent state.

SECONDARY OUTCOMES:
Patient's Glasgow Coma Scale (GCS) | According to the literature it is estimated to last approx. 70 days
  Calculation of GCS (range 0-15 with 15 being the normal) at the beginning and at the end of the CPM program.Until there is evidence by CT and laboratory measurements (bone Alkaline Phosphatase) that osteogenesis has entered a quiescent state.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical and Rehabilitation Medicine, Ioannina, Epirus, Greece

REFERENCES:
- [Background] Scalzitti DA. Because of the risk of developing heterotopic ossification, are passive range of motion exercises contraindicated following traumatic injuries? Phys Ther. 2003 Jul;83(7):659-7. No abstract available. PMID 12872776
- [Background] Vasileiadis GI, Varvarousis DN, Manolis I, Ploumis A. The Impact of Continuous Passive Motion on Heterotopic Ossification Maturation. Am J Phys Med Rehabil. 2021 Dec 1;100(12):e194-e197. doi: 10.1097/PHM.0000000000001852. PMID 34310347
- [Background] Vasileiadis GI, Balta AA, Zerva A, Kontogiannopoulos V, Varvarousis DN, Dimakopoulos G, Ploumis A. Role of Kinesiotherapy in the Prevention of Heterotopic Ossification: A Systematic Review. Am J Phys Med Rehabil. 2023 Feb 1;102(2):110-119. doi: 10.1097/PHM.0000000000002043. Epub 2022 Apr 28. PMID 35512120
- [Background] Genet F, Chehensse C, Jourdan C, Lautridou C, Denormandie P, Schnitzler A. Impact of the operative delay and the degree of neurologic sequelae on recurrence of excised heterotopic ossification in patients with traumatic brain injury. J Head Trauma Rehabil. 2012 Nov-Dec;27(6):443-8. doi: 10.1097/HTR.0b013e31822b54ba. PMID 22495100
- [Background] van Kampen PJ, Martina JD, Vos PE, Hoedemaekers CW, Hendricks HT. Potential risk factors for developing heterotopic ossification in patients with severe traumatic brain injury. J Head Trauma Rehabil. 2011 Sep-Oct;26(5):384-91. doi: 10.1097/HTR.0b013e3181f78a59. PMID 21321512
- [Background] Citak M, Suero EM, Backhaus M, Aach M, Godry H, Meindl R, Schildhauer TA. Risk factors for heterotopic ossification in patients with spinal cord injury: a case-control study of 264 patients. Spine (Phila Pa 1976). 2012 Nov 1;37(23):1953-7. doi: 10.1097/BRS.0b013e31825ee81b. PMID 22614800
- [Background] Shehab D, Elgazzar AH, Collier BD. Heterotopic ossification. J Nucl Med. 2002 Mar;43(3):346-53. PMID 11884494
- [Background] Holguin PH, Rico AA, Garcia JP, Del Rio JL. Elbow anchylosis due to postburn heterotopic ossification. J Burn Care Rehabil. 1996 Mar-Apr;17(2):150-4. doi: 10.1097/00004630-199603000-00009. PMID 8675505
- [Background] Linan E, O'Dell MW, Pierce JM. Continuous passive motion in the management of heterotopic ossification in a brain injured patient. Am J Phys Med Rehabil. 2001 Aug;80(8):614-7. doi: 10.1097/00002060-200108000-00013. PMID 11475483
- [Background] Stover SL, Hataway CJ, Zeiger HE. Heterotopic ossification in spinal cord-injured patients. Arch Phys Med Rehabil. 1975 May;56(5):199-204. PMID 806274